CLINICAL TRIAL: NCT07141589
Title: Fentanyl Versus Ketorolac as an Adjuvant to Peribulbar Block for Anterior Segment Surgeries, A Prospective Double-blinded Randomized Controlled Study
Brief Title: Fentanyl Versus Ketorolac as an Adjuvant to Peribulbar Block for Anterior Segment Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Abo Zied, Assistant Lecturer of Anesthesia, Surgical ICU and Pain Medicine, Faculty of Medicine, Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-264-2024
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Fentanyl; Ketorolac; Adjuvant; Peribulbar Block; Anterior Segment Surgeries
MeSH Terms: interventions — Lidocaine; Bupivacaine; Hyaluronoglucosaminidase; Fentanyl; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Patients will receive a mixture of 3 ml lidocaine 2%, 3 ml bupivacaine 0.5%, hyaluronidase 60 IU diluted in normal saline to a total volume of 8 ml.
  Interventions: Drug: Lidocaine + Bupivacaine + Hyaluronidase
- Fentanyl group (Experimental): Patients will receive a mixture of 3 ml lidocaine 2%, 3 ml bupivacaine 0.5%, and hyaluronidase 60 IU and fentanyl 20 μg diluted in normal saline to a total volume of 8 ml.
  Interventions: Drug: Fentanyl + Lidocaine + Bupivacaine + Hyaluronidase
- Ketorolac group (Experimental): Patients will receive a mixture of 3 ml lidocaine 2%, 3 ml bupivacaine 0.5%, hyaluronidase 60 IU, and ketorolac 15 mg diluted in normal saline to a total volume of 8 ml.
  Interventions: Drug: Ketorolac + Lidocaine + Bupivacaine + Hyaluronidase

INTERVENTIONS:
Drug: Lidocaine + Bupivacaine + Hyaluronidase — Patients will receive a mixture of 3 ml lidocaine 2%, 3 ml bupivacaine 0.5%, and hyaluronidase 60 IU diluted in normal saline to a total volume of 8 ml.
  Arms: Control group
Drug: Fentanyl + Lidocaine + Bupivacaine + Hyaluronidase — Patients will receive a mixture of 3 ml lidocaine 2%, 3 ml bupivacaine 0.5%, and hyaluronidase 60 IU and fentanyl 20 μg diluted in normal saline to a total volume of 8 ml.
  Arms: Fentanyl group
Drug: Ketorolac + Lidocaine + Bupivacaine + Hyaluronidase — Patients will receive a mixture of 3 ml lidocaine 2%, 3 ml bupivacaine 0.5%, hyaluronidase 60 IU, and ketorolac 15 mg diluted in normal saline to a total volume of 8 ml.
  Arms: Ketorolac group

SUMMARY:
This study aims to compare the efficacy of ketorolac and fentanyl as adjuvants to local anesthetics for anterior segment surgeries of the eye.

DETAILED DESCRIPTION:
Regional anesthesia for eye surgery includes peribulbar, retrobulbar, and sub-Tenon's blocks. Peribulbar block is commonly used due to a lesser incidence of serious complications such as globe perforation and retrobulbar hemorrhage.

Fentanyl is a synthetic opioid widely used as an adjuvant to local anesthetics to prolong its action and provide better postoperative analgesia. fentanyl fastens lid and globe akinesia and provides a better akinesia score.

Ketorolac is a non-steroidal anti-inflammatory drug (NSAID) that reduces the release of inflammatory mediators such as prostaglandins, thereby reducing afferent sensitivities and finally reducing pain. It is devoid of narcotic analgesic adverse effects such as sedation, nausea, and respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Scheduled to undergo operations for anterior segment surgeries of the eye under local (peribulbar) anesthesia.

Exclusion Criteria:

* Patient's refusal.
* Known allergy or hypersensitivity to aspirin or nonsteroidal anti-inflammatory medications.
* Patients with contraindications to local anesthetics, such as high axial length or patients with high preoperative intraocular pressure.
* If cases develop severe pain intraoperatively from the start, necessitating rescue analgesia and sedation or requiring conversion to general anesthesia.
* Infection at the site of injection.
* Patients with coagulopathies or on anticoagulants.
* Impaired renal function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Duration of globe akinesia | 10 minutes after injection
  Assessment of Globe akinesia will be assessed at 2, 5 and 10 minutes after injection with a 12-point scale. Each of the four rectus muscles and each lid score from 0 to 2; 0 = total akinesia, 1 = partial akinesia, 2 = no akinesia)

SECONDARY OUTCOMES:
Heart rate | Intraoperatively
  Intraoperative heart rate will be recorded every 5 minutes in beats per minute.
Blood pressure | Intraoperatively
  Intraoperative blood pressure will be recorded every 5 minutes in mmHg.
Onset of globe akinesia | 10 minutes after injection
  The onset of lid akinesia will be the elapsed time between the peribulbar injection and partial loss of lid movement.
Onset of corneal anesthesia | 1 minute after injection
  The onset of anesthesia will be defined as the time interval between performing the block and loss of corneal sensation.
Degree of pain | 6 hours postoperatively
  Pain will be assessed immediately after the operation , then after 1 h, 2 h, 4 h and 6 h by verbal rating scale (VRS) on a scale of 0-10 (where 0 no pain, and 10 worst imaginable pain).
Time of first rescue analgesia | 6 hours postoperatively
  Time of first rescue analgesia will be recorded from the end of surgery till first dose of opioid administrated.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.